CLINICAL TRIAL: NCT02412085
Title: Pilot Study to Evaluate the Efficacy of Golimumab for Induction and Maintenance of Clinical and Endoscopic Remission in Patients With Steroid-dependent Ulcerative Colitis
Brief Title: Golimumab in Steroid-dependent Ulcerative Colitis: Induction and Maintenance of Clinical and Endoscopic Remission
Acronym: UC-GOL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1371
Record Dates: First submitted 2015-03-26; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Colitis, Ulcerative
Keywords: golimumab; ulcerative colitis; steroid-dependent
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Golimumab (Experimental): Subcutaneous golimumab
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Subcutaneous golimumab. Induction regimen: 200 mg (week 0), 100 mg (week 2)
  Maintenance regimen:
  * body weight < 80kg: 50 mg every 4 weeks
  * body weight ≥ 80 kg: 100 mg every 4 weeks
  Other Names: Simponi

SUMMARY:
This is an open-label, phase IV trial. Adult patients, with moderately to severe, steroid dependent, acute ulcerative colitis not previously exposed to anti-TNF, will receive subcutaneous golimumab treatment, according to EU marketing authorization from baseline through week 14.

At week 16, patients achieving clinical and endoscopic remission will continue with Golimumab, 50 mg or 100 mg (depending on body weight) every 4 weeks, through week 52.

Patients not achieving clinical and endoscopic remission will be treated with infliximab, according to marketing authorization, and followed through week 52. This is not considered as an interventional arm but, since infliximab in Italy is considered as the first-line treatment for UC patients, as the usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65 years
* ability to understand the study procedures and sign the informed consent
* ulcerative colitis diagnosed at least 6 months before
* no previous exposure to anti-TNFs
* Global Mayo score ≥ 6 (with endoscopic sub-score ≥2) at baseline
* steroid-dependent disease
* women of childbearing potential must accept effective contraception during study participation and for at leas 6 months after the end of study participation

Exclusion Criteria:

* Crohn's disease or undetermined colitis
* active infections or previous infections not completely resolved at baseline
* malignancies in the previous 5 years
* suspected latent tuberculosis infection
* every other potentially harmful clinical condition, in the opinion of the investigator
* patients with moderately to severe heart failure (NYHA class III/IV)
* hepatic or renal failure
* pregnant or lactating women or women planning a pregnancy between baseline and the 3 months after study completion
* not permitted concomitant medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
clinical and endoscopic steroid-free remission | week 16
  Total Mayo score ≤2, with no sub-score >1. No concomitant corticosteroid therapy.

SECONDARY OUTCOMES:
clinical response | week 16
  Decrease in total Mayo score of at least 2 point and 30 %
percentage of patients in clinical and endoscopic remission | week 52
  Total Mayo score ≤2, with no sub-score >1
percentage of patients in clinical remission | week 52
  partial Mayo score ≤2, with no sub-score >1
percentage of patients with mucosal healing | week 16 and 52
  complete mucosal healing: endoscopic sub-score 0
percentage of patients with histological healing | week 16 and 52
  histological healing: Geboes score <3 and no Mayo sub-score >1
quality of life | week 16 and 52
  IBDQ questionnaire
percentage of infliximab responders | week 52
identification of patients that would benefit from golimumab therapy | through week 52
  evaluation of baseline characteristics of patients to identify potential response-predictive factors.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, MD, PhD, Study Chair — IBD Center, Humanitas Research Hospital, Rozzano (MI) ITALY
Locations (1):
- IBD Center, Rozzano, MI, Italy